CLINICAL TRIAL: NCT05663138
Title: The Outcome of Early Use of High-velocity Nasal Insufflation in Acute Respiratory Failure Complicating Covid-19
Brief Title: Early Versus Late Use of Hi-VNI in Covid-19
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Aswan University (Other)
Responsible Party: Principal Investigator, Lamees Mohamed Bakkar, clinical professor, Assiut University
Other Study IDs: Hi-VNI in covid 19 patients
Record Dates: First submitted 2022-12-20; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Hi-VNI; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Hi-VNI: Group 1 of early shift to Hi-VNI after nasal cannula
- Late Hi-VNI: Group 2 of late use of Hi-VNI after NRM

SUMMARY:
This study evaluate early administration of high-velocity nasal insufflation in COVID-19 patients presented with acute respiratory failure after failure of conventional low flow nasal cannula bypassing the escalating step of Non re-breathing mask where early use of High velocity nasal insufflations achieved better improvement of respiratory distress, lower oxygen requirements and shorter ICU stay.

DETAILED DESCRIPTION:
The study included 30 COVID-19 patients admitted to intensive care of COVID-19 zone, chest Department, quarantine section, Assiut University hospital. All patients were positive for COVID-19 infection by nasopharyngeal swab for detection of viral RNA by real time PCR for SAR-COV-2 RNA assay on 7500 Applied Bio-system. All patients received treatment based on the protocol of Egyptian Ministry of Health, Patients enrolled in the study were categorized into 2 groups, the 1st group included patients whom were shifted to Hi-VNI after failure of high flow nasal cannula, while the 2nd group included patients shifted to Hi-VNI after failure of non-rebreathing mask, using a Precision flow vapotherm (vapotherm, Inc, 100 Domain device Exeter, NH 03833, T: 603-658-0011, USA), that provide high velocity humidified flow through narrow bore nasl prongs

ELIGIBILITY:
Inclusion Criteria:

* 1-severe COVID Patients with hypoxemic respiratory failure. 2- Patients with no comorbidities

Exclusion Criteria:

1. Non severe COVID Patients
2. Patients with comorbidities (e.g chronic chest dis, DM, renal failure and hepatic failure
3. Patients indicated for mechanical ventilation
4. Patients with marked hypercapnia in need for non-invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as COVID-19 presented with respiratory failure and admitted to intensive care of COVID-19 zone, chest Department, Assiut University hospital, Patients who failed on either low flow nasal cannula or non-rebreathing mask were shifted to Hi-VNI device using a Precision flow vapotherm (vapotherm, Inc, 100 Domain device Exeter, NH 03833, T: 603-658-0011, USA). Patients were classified into 2 groups: Early and late Hi-VNI groups according to whether the shift to Hi-VNI occurred after low flow nasal cannula or non-rebreathing mask respectively.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Improved oxygenation | through the study completion, average 6 months
  Patients with early use of Hi-VNI had better improvement of oxygenation than those with late use of Hi-VNI

CONTACTS AND LOCATIONS:
Overall Officials: Lamees M Bakkar, Fellow, Principal Investigator — Fellow of Chest diseases Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granton D, Chaudhuri D, Wang D, Einav S, Helviz Y, Mauri T, Mancebo J, Frat JP, Jog S, Hernandez G, Maggiore SM, Hodgson CL, Jaber S, Brochard L, Trivedi V, Ricard JD, Goligher EC, Burns KEA, Rochwerg B. High-Flow Nasal Cannula Compared With Conventional Oxygen Therapy or Noninvasive Ventilation Immediately Postextubation: A Systematic Review and Meta-Analysis. Crit Care Med. 2020 Nov;48(11):e1129-e1136. doi: 10.1097/CCM.0000000000004576. PMID 32947472
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464